CLINICAL TRIAL: NCT05798884
Title: Electro-acupuncture for the Prevention and Treatment of Oxaliplatin-induced Neurotoxicity in Colorectal Cancer Patients: a Prospective, Randomized, Sham-controlled, Double-blinded and Multicenter Study
Brief Title: Electro-acupuncture for the Prevention and Treatment of Oxaliplatin-induced Neurotoxicity in Colorectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government); Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020HMRF
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Oxaliplatin; Electro-acupuncture; Neurotoxicity
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All patients and the investigators including the research assessors, the statistician, and the researchers interacting with the patients except the one who conducts the acupuncture therapy will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture group (Experimental): The electro-acupuncture intervention will be conducted for 2 sessions per week for 4 consecutive weeks before and 8 weeks during the chemotherapy. In this study eight acupoints are chosen: he gu (LI4), nei guan (PC6), qu chi (LI12), ba xie (EX-UE9), zu san li (ST36), san yin jiao (SP6), tai chung (LV3) and ba feng (EX-LE10). The use of ba xie (EX-UE9) and ba feng (EX-LE10) will be optional if skin lesions of hands and feet occur due to Capecitabine (Xeloda). Disposable acupuncture needles (verum acupuncture needles Hwato 0.25 x 25mm matching the Streiterger sham needles) will be inserted at a depth of 10-25mm into the points. Electrical stimulation will be delivered with continuous waves at 2 Hz, at an intensity of each patient's minimum sensation of stimulation through the electrical acupuncture stimulation instrument. The needles will be retained in position for 25 minutes.
  Interventions: Device: Acupuncture
- sham-acupuncture group (Sham Comparator): For subjects assigned to the sham control group, Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2"/ 0.30 x 30mm) will be applied to serve as a sham control at the same acupoints with the same stimulation modality, and the stimulation will be a "pseudo stimulation", which will be given by connecting the needle to the incorrect output socket of the electrical acupuncture stimulation instrument.The credibility and validity of this system have been well demonstrated.
  Interventions: Device: Sham-acupuncture

INTERVENTIONS:
Device: Acupuncture — Disposable acupuncture needles (0.25 mm in diameter and 25 mm in length) are straightly into body acupuncture points (he gu (LI4), nei guan (PC6), qu chi (LI12), ba xie (EX-UE9), zu san li (ST36), san yin jiao (SP6), tai chung (LV3) and ba feng (EX-LE10)). The use of ba xie (EX-UE9) and ba feng (EX-LE10) will be optional if skin lesions of hands and feet occur due to Capecitabine (Xeloda). Electrical stimulation will be delivered with continuous waves at 2 Hz, at an intensity of each patient's minimum sensation of stimulation through the electrical acupuncture stimulation instrument. The needles will be retained in position for 25 minutes.
  Arms: Electro-acupuncture group
Device: Sham-acupuncture — Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2"/ 0.30 x 30mm) will be applied to serve as a sham control at the same acupoints with the same stimulation modality and then connecting the needle to the incorrect output socket of the electrical acupuncture stimulation instrument. The sham points are "pseudo stimulation".
  Arms: sham-acupuncture group

SUMMARY:
In this study, a 24-week randomized, sham-controlled, single-blind, multicenter clinical trial will be conducted to explore the effect of electroacupuncture for prevention and treatment of both acute and chronic neurotoxicity through both clinical and biological indicators.

DETAILED DESCRIPTION:
This is a prospective, randomized, sham-controlled, double-blinded and multiple center trial on electro-acupuncture for preventing and treating symptoms of chemotherapy-induced neurotoxicity in patients with colorectal cancer. A total of 150 candidates will be recruited in this study four weeks before chemotherapy for best preventive effect. They will be assigned randomly into either the electro-acupuncture or the sham-control group with 1:1 ratio. Both groups will receive a total of 24 sessions of interventions (4 weeks before chemotherapy and 8 weeks during chemotherapy, with 2 session per week), and will be followed up regularly for up to 12 weeks after completion of the acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* are aged ≥18 years old;
* are newly diagnosed with stage II to IV colorectal cancer;
* going to receive adjuvant oxaliplatin-based chemotherapy within 4 weeks;
* had not received any acupuncture in the previous 3 months and had a life expectancy ≥ of six months.

Exclusion Criteria:

* are not able to comprehend and communicate;
* are not able to read Chinese;
* have prior peripheral neuropathy caused by other diseases including diabetes, stroke, cardiovascular diseases such as arrhythmia, heart failure, myocardial infarction, and patients with cardiac pacemakers;
* have a bleeding tendency;
* are pregnant or breastfeeding;
* have impaired hepatic or renal function;
* using any pharmaceutical agents e.g., vitamin B6 and vitamin E, or herbal medication. All the above medication prescribed by physicians or Chinese medicine practitioners during the study will be recorded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Score Changes on the FACT/GOG-Ntx questionnaire | 0-24 weeks; weekly
  The questionnaire includes 11 questions covering sensory neuropathy, motor neuropathy, hearing neuropathy, and dysfunction associated with neuropathy, which results in a cumulative score ranging from 0 to 44, with the lower scores reflecting worse neuropathy symptoms.

SECONDARY OUTCOMES:
numerical rating scale (NRS) | 0-24 weeks; weekly
  Patients will be asked to rate their average neuropathy symptoms within one week, on an 0 to 10 scale (0=no symptoms; 10=worst possible symptoms), those <4 of 10 NRS will be considered as mild neuropathy while ≥4 of 10 NRS will be considered as moderate to severe neuropathy.
European Organization for Research and Treatment of Cancer (EORCTC) quality of life questionnaire QLQ-C30 | 0,3,6,9,12,15,18,21,24 weeks
  A 30-items questionnaire assessing five functional scales (physical, role, cognitive, emotional and social), three symptoms scales (fatigue, pain, nausea and vomiting), and other symptoms and problem in cancer patients (dyspnoea, appetite loss, insomnia, constipation, diarrhoea, and financial difficulties).
Constitution of Chinese Medicine Questionnaire (CCMQ) | 0,12,24 weeks
  CCMQ has 60 items measuring the 9 body constitution types: gentleness, Qi-deficiency, Yang-deficiency, Yin-deficiency, phlegm-wetness, wetness-heat, blood-stasis, Qi-depression, and special diathesis.
Vibration sense test | 0-12 week; weekly
  It will be assessed using the graduated Rydel-Seiffer tuning fork (U.S. Neurologicals, Poulsbo, WA), with printed directions for use and its normative data. Readings will be averaged and recorded as the vibration value.
Light touch test | 0-12 week; weekly
  It will be assessed with standard 10g monofilaments, contained within the Neuropen (Owen Mumford, Woodstock, UK). During testing, the fiber will be applied perpendicular to the plantar surface of the great toe and the palmar surface of the index finger until the fiber begins to bend and will be held in place for 1 second and then removed. This procedure will be repeated 3 times and the patient will be asked to report the ability to feel the fibe.
Short Form 12 item(version 2) Health Survey (SF-12V2) | 0-12 week; weekly
  The SF-12V2 is a widely used generic HRQoL instrument, and its Chinese version has been validated and normed in the general Chinese population in Hong Kong. It consists of 12 questions measuring eight domains of health, including physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The scores are generated using an algorithm to generate a combined physical and mental health score for comparison with normative data. In the normative data: 1) the mean score was set to 50; 2) a score > 50 indicated better physical or mental health than the mean; 3) a score < 50 indicated worse physical or mental health than the mean.

CONTACTS AND LOCATIONS:
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hospital Authority. Hong Kong Cancer Registry. https://www3.ha.org.hk/cancereg/ (accessed on 29 March 2021)
- [Background] Engstrom PF, Arnoletti JP, Benson AB 3rd, Chen YJ, Choti MA, Cooper HS, Covey A, Dilawari RA, Early DS, Enzinger PC, Fakih MG, Fleshman J Jr, Fuchs C, Grem JL, Kiel K, Knol JA, Leong LA, Lin E, Mulcahy MF, Rao S, Ryan DP, Saltz L, Shibata D, Skibber JM, Sofocleous C, Thomas J, Venook AP, Willett C; National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: colon cancer. J Natl Compr Canc Netw. 2009 Sep;7(8):778-831. doi: 10.6004/jnccn.2009.0056. No abstract available. PMID 19755046
- [Background] Tofthagen C, Donovan KA, Morgan MA, Shibata D, Yeh Y. Oxaliplatin-induced peripheral neuropathy's effects on health-related quality of life of colorectal cancer survivors. Support Care Cancer. 2013 Dec;21(12):3307-13. doi: 10.1007/s00520-013-1905-5. Epub 2013 Aug 1. PMID 23903798
- [Background] Sato J, Mori M, Nihei S, Takeuchi S, Kashiwaba M, Kudo K. Objective evaluation of chemotherapy-induced peripheral neuropathy using quantitative pain measurement system (Pain Vision(R)), a pilot study. J Pharm Health Care Sci. 2017 Jul 25;3:21. doi: 10.1186/s40780-017-0089-4. eCollection 2017. PMID 28770097
- [Background] Wang X, Wei G, Huo J. Chinese medicine for prevention and treatment of oxaliplatin-induced peripheral neuropathy. Jilin J Chinese Med 2013; 5: 465-467.
- [Background] Brami C, Bao T, Deng G. Natural products and complementary therapies for chemotherapy-induced peripheral neuropathy: A systematic review. Crit Rev Oncol Hematol. 2016 Feb;98:325-34. doi: 10.1016/j.critrevonc.2015.11.014. Epub 2015 Nov 23. PMID 26652982
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Greenlee H, Crew KD, Capodice J, Awad D, Buono D, Shi Z, Jeffres A, Wyse S, Whitman W, Trivedi MS, Kalinsky K, Hershman DL. Randomized sham-controlled pilot trial of weekly electro-acupuncture for the prevention of taxane-induced peripheral neuropathy in women with early stage breast cancer. Breast Cancer Res Treat. 2016 Apr;156(3):453-464. doi: 10.1007/s10549-016-3759-2. Epub 2016 Mar 25. PMID 27013473
- [Background] Han X, Wang L, Shi H, Zheng G, He J, Wu W, Shi J, Wei G, Zheng W, Sun J, Huang H, Cai Z. Acupuncture combined with methylcobalamin for the treatment of chemotherapy-induced peripheral neuropathy in patients with multiple myeloma. BMC Cancer. 2017 Jan 9;17(1):40. doi: 10.1186/s12885-016-3037-z. PMID 28068938
- [Background] Rostock M, Jaroslawski K, Guethlin C, Ludtke R, Schroder S, Bartsch HH. Chemotherapy-induced peripheral neuropathy in cancer patients: a four-arm randomized trial on the effectiveness of electroacupuncture. Evid Based Complement Alternat Med. 2013;2013:349653. doi: 10.1155/2013/349653. Epub 2013 Aug 28. PMID 24066010
- [Background] Derksen TM, Bours MJ, Mols F, Weijenberg MP. Lifestyle-Related Factors in the Self-Management of Chemotherapy-Induced Peripheral Neuropathy in Colorectal Cancer: A Systematic Review. Evid Based Complement Alternat Med. 2017;2017:7916031. doi: 10.1155/2017/7916031. Epub 2017 Mar 16. PMID 28400846
- [Background] Chan K, Lui L, Yu K, Lau K, Lai M, Lau W, Ng B, Zhong LLD, Bian ZX. The efficacy and safety of electro-acupuncture for alleviating chemotherapy-induced peripheral neuropathy in patients with coloreactal cancer: study protocol for a single-blinded, randomized sham-controlled trial. Trials. 2020 Jan 9;21(1):58. doi: 10.1186/s13063-019-3972-5. PMID 31918748
- [Background] Lu Z, Moody J, Marx BL, Hammerstrom T. Treatment of Chemotherapy-Induced Peripheral Neuropathy in Integrative Oncology: A Survey of Acupuncture and Oriental Medicine Practitioners. J Altern Complement Med. 2017 Dec;23(12):964-970. doi: 10.1089/acm.2017.0052. Epub 2017 Jun 29. PMID 28661695
- [Background] Shin KM, Kim JH, Lee S, Shin MS, Kim TH, Park HJ, Lee MH, Hong KE, Lee S, Choi SM. Acupuncture for lateral epicondylitis (tennis elbow): study protocol for a randomized, practitioner-assessor blinded, controlled pilot clinical trial. Trials. 2013 Jun 14;14:174. doi: 10.1186/1745-6215-14-174. PMID 23768129
- [Background] Xie CC, Wen XY, Jiang L, Xie MJ, Fu WB. Validity of the "streitberger" needle in a chinese population with acupuncture: a randomized, single-blinded, and crossover pilot study. Evid Based Complement Alternat Med. 2013;2013:251603. doi: 10.1155/2013/251603. Epub 2013 Aug 1. PMID 23983775
- [Background] Fleckenstein J, Baeumler PI, Gurschler C, Weissenbacher T, Simang M, Annecke T, Geisenberger T, Irnich D. Acupuncture for post anaesthetic recovery and postoperative pain: study protocol for a randomised controlled trial. Trials. 2014 Jul 21;15:292. doi: 10.1186/1745-6215-15-292. PMID 25047046
- [Background] Man SC, Hung BH, Ng RM, Yu XC, Cheung H, Fung MP, Li LS, Leung KP, Leung KP, Tsang KW, Ziea E, Wong VT, Zhang ZJ. A pilot controlled trial of a combination of dense cranial electroacupuncture stimulation and body acupuncture for post-stroke depression. BMC Complement Altern Med. 2014 Jul 19;14:255. doi: 10.1186/1472-6882-14-255. PMID 25038733
- [Background] Huang HQ, Brady MF, Cella D, Fleming G. Validation and reduction of FACT/GOG-Ntx subscale for platinum/paclitaxel-induced neurologic symptoms: a gynecologic oncology group study. Int J Gynecol Cancer. 2007 Mar-Apr;17(2):387-93. doi: 10.1111/j.1525-1438.2007.00794.x. PMID 17362317
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309
- [Background] Gewandter JS, Dworkin RH, Finnerup NB, Mohile NA. Painful chemotherapy-induced peripheral neuropathy: lack of treatment efficacy or the wrong clinical trial methodology? Pain. 2017 Jan;158(1):30-33. doi: 10.1097/j.pain.0000000000000653. No abstract available. PMID 27564867
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Wong W, Lam CL, Wong VT, Yang ZM, Ziea ET, Kwan AK. Validation of the constitution in chinese medicine questionnaire: does the traditional chinese medicine concept of body constitution exist? Evid Based Complement Alternat Med. 2013;2013:481491. doi: 10.1155/2013/481491. Epub 2013 Apr 24. PMID 23710222
- [Background] Wong W, Lam CL, Su YC, Lin SJ, Ziea ET, Wong VT, Wai LK, Kwan AK. Measuring body constitution: validation of the Body Constitution Questionnaire (BCQ) in Hong Kong. Complement Ther Med. 2014 Aug;22(4):670-82. doi: 10.1016/j.ctim.2014.05.009. Epub 2014 May 27. PMID 25146072
- [Background] Griffith KA, Dorsey SG, Renn CL, Zhu S, Johantgen ME, Cornblath DR, Argyriou AA, Cavaletti G, Merkies IS, Alberti P, Postma TJ, Rossi E, Frigeni B, Bruna J, Velasco R, Kalofonos HP, Psimaras D, Ricard D, Pace A, Galie E, Briani C, Dalla Torre C, Faber CG, Lalisang RI, Boogerd W, Brandsma D, Koeppen S, Hense J, Storey DJ, Kerrigan S, Schenone A, Fabbri S, Valsecchi MG; CI-PeriNomS Group. Correspondence between neurophysiological and clinical measurements of chemotherapy-induced peripheral neuropathy: secondary analysis of data from the CI-PeriNomS study. J Peripher Nerv Syst. 2014 Jun;19(2):127-35. doi: 10.1111/jns5.12064. PMID 24814100
- [Background] El-Fatatry BM, Ibrahim OM, Hussien FZ, Mostafa TM. Role of metformin in oxaliplatin-induced peripheral neuropathy in patients with stage III colorectal cancer: randomized, controlled study. Int J Colorectal Dis. 2018 Dec;33(12):1675-1683. doi: 10.1007/s00384-018-3104-9. Epub 2018 Jun 21. PMID 29931409
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- See also: accessed on 29 March 2021 — https://www3.ha.org.hk/cancereg/